CLINICAL TRIAL: NCT02781363
Title: Can the Thoracic Replace the Conventional Radiography for the Diagnosis of Acute Pneumonia in Children?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The principal investigator left the center in 2016.
Sponsor: Hospital Universitari General de Catalunya (Other)
Responsible Party: Principal Investigator, Montse Granados, Hospital Universitari General de Catalunya, Hospital Universitari General de Catalunya
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2015/51-PED-HGC
Record Dates: First submitted 2016-05-18; First posted 2016-05-24 (Estimated); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Pneumonia
Keywords: thoracic ultrasound; children; efficacy; emergency service
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Candidates patients chest X-ray with pneumonia (Other): thoracic sonography CXR Clinical control 48h
  Interventions: Other: Thoracic ultrasound; Other: CXR
- Candidates patients chest X-ray without pneumonia (Other): thoracic sonography CXR Clinical control 48h
  Interventions: Other: Thoracic ultrasound; Other: CXR

INTERVENTIONS:
Other: Thoracic ultrasound
Other: CXR

SUMMARY:
The Thoracic ultrasound is a safer and sensitive technique than conventional radiography because it detects less than 1 cm pneumonic consolidations and minimal pleural effusions. The main objective is to evaluate the efficacy of thoracic ultrasound performed by unskilled personnel in the emergency service prdiatricas to diagnose pneumonia in children.

DETAILED DESCRIPTION:
Diagnostic test evaluation.The sample collected sequentially until an exact size . Given the safety of the technique, which involves no risk to patient management and the possibility of generating a type II error by premature study discontinuation , we have no plans to make any interim analyzes .

ELIGIBILITY:
Inclusion Criteria:

* fever above 38 degrees
* tachypnea
* Difficulty breathing
* Side tip pain
* pathological auscultation

Exclusion Criteria:

* < 3 months> 14 years
* Background of Prematurity
* Rewalizados imaging studies in the last 7 days
* Any chronic respiratory process
* congenital heart diseases
* hemodynamic instability
* Diagnosis of pneumonia in the last 3 months
* Refusal of relatives to participate in the study

Ages: 3 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
coincidence between the ultrasound image and conventional radiography | 1 day
  images compatible with pneumonic consolidations in sonography and radiography . Coincidence between evaluators

SECONDARY OUTCOMES:
additional workload | 1 day
  Time (minutes) between the test requested and the results are obtained for both diagnostic tests

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital UNiversitari General de Catalunya, Sant Cugat del Vallès, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No